CLINICAL TRIAL: NCT07333599
Title: Hypoxia Profiles Identified in Term Newborns With Cord pH <7.00
Acronym: RCFHypA
Status: Recruiting | Type: Observational
Sponsor: University Hospital, Strasbourg, France (Other)
Responsible Party: Sponsor
Other Study IDs: 9618
Record Dates: First submitted 2025-12-31; First posted 2026-01-12 (Actual); Last update posted 2026-01-12 (Actual); Status verified 2025-12

CONDITIONS: Neonatal Acidemia and Hypoxia
Keywords: Hypoxia Neonatal; Neonatal acidosis; Neonatal Acidemia; Obstetrical Surgery; Newborns
MeSH Terms: conditions — Hypoxia; Asphyxia Neonatorum

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Severe neonatal acidosis is an identified risk factor for neonatal encephalopathies and severe neurological sequelae such as cerebral palsy. While intrapartum origin of such deterioration is rare (approximately 20% of adverse outcomes in term infants), screening for hypoxia that can lead to the development of severe acidosis remains inadequate. This results in both delays in diagnosis and/or intervention, and a parallel increase in obstetric interventions (cesarean sections and operative vaginal deliveries) sometimes performed with inappropriate indications, thus contributing to unnecessary maternal and neonatal comorbidities. Difficulties in analyzing fetal heart rate (FHR) patterns are identified as an independent risk factor, particularly due to significant inter- and intra-observer variability, in an examination that is nevertheless central to assessing fetal well-being during labor. An FHR analysis based on a thorough understanding of the physiology of fetal adaptation to hypoxia could allow for better recognition of situations where fetal compensation for hypoxic stress is no longer possible, when adaptive mechanisms are exhausted. Given that FHR interpretation errors are implicated in 35 to 50% of adverse neonatal outcomes (peripartum death, early neonatal death, or irreversible brain damage), the preventability of these traumatic complications for families is systematically called into question. Furthermore, recent data suggest that defining hypoxia profiles associated with tracing characteristics would allow for more accurate identification of these situations, and for improved use of intervention in a more appropriate manner in terms of time and resources, in an attempt to reduce the incidence of neonatal complications of hypoxic origin involved in the development of severe neurological sequelae.

ELIGIBILITY:
Inclusion Criteria:

* Adult woman (≥ 18 years)
* Treated at Strasbourg University Hospital between January 1, 2014, and December 31, 2024
* Singleton pregnancy
* Cord arterial pH < 7.00

Exclusion Criteria:

* Gestational age < 37 weeks
* Known congenital malformation
* Intrauterine fetal death diagnosed upon admission
* No cardiotocographic recording

Ages: 0 Days to 1 Day | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Adult woman (≥ 18 years) with singleton pregnancy and cord arterial pH < 7.00
Sampling Method: Non-Probability Sample
Enrollment: 400 (Estimated)
Dates: Start 2025-04-04 (Actual); Primary Completion 2026-08 (Estimated); Study Completion 2026-08-14 (Estimated)

PRIMARY OUTCOMES:
Apgar score | The score is measured 1 minute and 5 minutes after birth.
  Apgar score:
  * 7 to 10 points: Healthy baby
  * 4 to 6 points: The baby needs some help (oxygen, stimulation, etc.)
  * 0 to 3 points: Urgent situation; the baby needs immediate care

CONTACTS AND LOCATIONS:
Locations (1):
- Service de Gynécologie-Obstétrique - CHU de Strasbourg - France, Strasbourg, France